CLINICAL TRIAL: NCT03708666
Title: Nephrocare mHealth: Improvement of Patient Empowerment and Self-management by the Use of Telemonitoring.
Brief Title: Nephrocare mHealth Project: Telemonitoring of Blood Pressure
Acronym: Nephrocare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Kathleen Claes, Prof. Dr. K. Claes, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S60335; AZGS2017056 (Other: AZ Groeninge)
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Diseases; Blood Pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telemonitoring of blood pressure (Other): Patients measure their blood pressure and register their results on the app or website.
  Interventions: Other: Telemonitoring of blood pressure

INTERVENTIONS:
Other: Telemonitoring of blood pressure — Blood pressure monitoring at least once a week.

SUMMARY:
The Nephrocare mHealth project supports patients with Chronic Kidney Disease with a mobile application and telemonitoring. The application includes the follow-up of blood pressure.

DETAILED DESCRIPTION:
Patients that are included in the Nephrocare mHealth project send their blood pressure results through an app or online website.

The clinical decision support system will alert the patient, as well as the general practitioner and the hospital when the blood pressure is too high or low. In addition the clinical decision support will calculate monthly averages and all the data are connected with the electronic patient files.

ELIGIBILITY:
Inclusion Criteria:

* Dutch-speaking
* Signed and approved informed consent
* Follow-up by nephrology at the University Hospitals Leuven or General Hospital Groeninge

Exclusion Criteria:

* No Dutch-speaking
* Impaired cognitive condition or medically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure under control | 6 months
  Percentage of patients with blood pressure within target limits

SECONDARY OUTCOMES:
Adaptations of treatment | 6 months
  Percentage of change in hypertension therapy

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Claes, Prof. Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No